CLINICAL TRIAL: NCT02143570
Title: Efficacy of Darifenacin and Physiotherapy for the Treatment of Overactive Bladder in Women
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Universidad de Valparaiso (Other)
Collaborators: Recalcine (GynoPharm) (Unknown)
Responsible Party: Principal Investigator, Felipe Martinez, M.D., M.Sc., Universidad de Valparaiso
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 635
Record Dates: First submitted 2014-05-18; First posted 2014-05-21 (Estimated); Last update posted 2016-05-02 (Estimated); Status verified 2016-04

CONDITIONS: Overactive Bladder
Keywords: Urinary Bladder, Overactive; Darifenacin; Physiotherapy; Quality of Life
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — darifenacin; Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Darifenacin + Physiotherapy (Experimental): Patients allocated to this group will receive Darifenacin 7.5mg daily in addition to physiotherapy for 12 weeks. This dose may be increased up to 7.5mg twice daily in follow-up visits in cases of refractory symptoms.
  Interventions: Drug: Darifenacin; Procedure: Physiotherapy
- Physiotherapy (Active Comparator): Patients allocated to this arm will receive a tailored pelvic floor exercise programme in addition to a matching placebo pill.
  Interventions: Procedure: Physiotherapy

INTERVENTIONS:
Drug: Darifenacin — Darifenacin will be prescribed in a starting dose of 7.5mg, once daily. This dose may be increased to 15mg a day in cases with refractory symptoms.
  Other Names: Oralafi; Darisec; Continex; Emselex; Enablex
  Arms: Darifenacin + Physiotherapy
Procedure: Physiotherapy — All patients will received a tailored pelvic floor exercise programme as part of the standard of care of overactive bladder at the study centre. This intervention will be mainly comprised of biofeedback stimulation techniques.

SUMMARY:
Overactive bladder is a common problem among adult women. Darifenacin is an antimuscarinic drug that is frequently used as part of the management of the condition. However, current evidence backing its use is limited. This study aims to address Darifenacin's effectiveness in adjunct to physiotherapy in treating symptoms due to overactive bladder.

ELIGIBILITY:
Inclusion Criteria:

* Patients with overactive bladder as diagnosed and confirmed by a urologist.
* Able to answer the ICIC, King's Health Questionnaire and Overactive Bladder Questionnaire.
* Able and willing to receive urodynamic studies.

Exclusion Criteria:

* History of pelvic radiotherapy.
* Recent pelvic surgery (<1 year).
* History of anti-incontinence surgery.
* Pregnancy.

Min Age: 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2014-05; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Quality of Life | 12 weeks
  Overall quality of life as established by the Overactive Bladder Questionnaire.

SECONDARY OUTCOMES:
Overactive Bladder Symptoms | 12 weeks
  Presence of symptoms of overactive bladder, as established by the King's Health Questionnaire and the International Consultation on Incontinence Questionnaire.
Adverse Events | 12 weeks
  Development of any adverse event attributable to darifenacin and as established by a standardised questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Cifuentes, M.D., Principal Investigator — Senior Urologist
Locations (1):
- Hospital Carlos Van Buren, Valparaíso, Región de Valparaíso, Chile

REFERENCES:
- [Derived] Stoniute A, Madhuvrata P, Still M, Barron-Millar E, Nabi G, Omar MI. Oral anticholinergic drugs versus placebo or no treatment for managing overactive bladder syndrome in adults. Cochrane Database Syst Rev. 2023 May 9;5(5):CD003781. doi: 10.1002/14651858.CD003781.pub3. PMID 37160401